CLINICAL TRIAL: NCT01913132
Title: PICO Versus Standard Dressing on Groin Incisions After Vascular Surgery - a Prospective Randomized Trial (INVIPS Trial)
Brief Title: PICO Above Incisions After Vascular Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefan Acosta (Other)
Responsible Party: Sponsor-Investigator, Stefan Acosta, Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr 2013/322
Record Dates: First submitted 2013-07-25; First posted 2013-07-31 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Wound; Infection
Keywords: Negative pressure wound therapy; Vascular Surgery; Inguinal incisions
MeSH Terms: conditions — Wounds and Injuries; Infections | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: 2 study subgroups: 1) OPEN arm for open procedures 2) EVAR arm for endovascular aortic repair
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard wound dressing OPEN (No Intervention): Standard wound dressing
- PICO dressing OPEN (Experimental): Negative pressure wound therapy with PICO (Smith & Nephew)
  Interventions: Device: Negative pressure wound therapy with PICO (Smith & Nephew)
- Standard dressing EVAR (No Intervention): Standard wound dressing
- PICO dressing EVAR (Experimental): Negative pressure wound therapy with PICO (Smith & Nephew)
  Interventions: Device: Negative pressure wound therapy with PICO (Smith & Nephew)

INTERVENTIONS:
Device: Negative pressure wound therapy with PICO (Smith & Nephew) — Negative wound pressure therapy
  Arms: PICO dressing EVAR; PICO dressing OPEN

SUMMARY:
The wound infection rate in the groin after vascular surgery has been denoted to be high since the wound surveillance register started in 2005. The current wound infection rate based on a validation study was 22.9% (24/105 patients with groin incision(s) between 1 March to 30 June in 2012). This randomized controlled trial aims to evaluate if negative pressure wound therapy on closed inguinal incisions (INPWT) after vascular surgical procedures can reduce the risk for surgical site infections and other wound complications.

DETAILED DESCRIPTION:
As published in the study´s rational and design paper (DOI: 10.4236/ss.2015.612080), we conducted a reanalysis of the material that the original power calculation was based on and included elective cases only which led to a slightly different number of cases needed. Furthermore, it became clear that there were big differences in the infection rates of EVAR (endovascular aortic repair) and open vascular procedures and therefore the need to split the study into two arms, an EVAR arm and an OPEN arm.

To prove a significant effect of the treatment intervention in the EVAR arm with a wound infection rate reduction from previously 4.4% to 1%, 80% power, 5% significance level and Including a margin for loss to follow-up, the EVAR arm requires 497 inguinal incisions. Assuming a surgical site infection rate reduction from 30% to 10% in the OPEN arm of the study, 80% power and 5% significance level, a total of 147 inguinal incisions is required.

We conducted an unannounced interim analysis for a conference presentation that was conducted by the study's principal investigators Stefan Acosta and Julien Hasselmann. Staff in charge of the day-to-day activities of the trial were not involved or actively informed of this. We believe that using an objective wound assessment tool (ASEPSIS score) minimizes any potential bias associated with the interim analysis.

Since the vascular center Malmö has started using closure-devices for almost all EVAR cases and thereby creating virtually no wounds to assess, we have started a multi center extension of the EVAR arm to Örebro University Hospital to be able to include the outstanding cases.

FUNDING

The trial has been funded by public Swedish funds stemming from the Southmost region in Sweden (Region Skåne), the Skåne University Hospital and the Hulda Almroth foundation since 2015 and adds up to a total of 2.81 million SEK (about 311,000 USD). In addition the research group received an unrestricted unconditional research grant of 15,550 USD and a donation of 100 PICO dressing kits from Smith and Nephew in 2013.

ALF (Agreement on medical education and research) funding has been granted for the time period 2019 - 2022 but has not yet been defined monetarily.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and above
* Elective vascular surgery
* Inguinal incision (transverse or longitudinal)
* Capable of understanding the study information and giving written informed consent

Exclusion Criteria:

* Emergency surgery
* Ongoing infection in inguinal area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wound infection rate | Wounds will be checked at 3 month follow-up
  ASEPSIS (Additional treatment, the presence of Serous discharge, Erythema, Purulent exudate, and Separation of the Deep tissues, the isolation of bacteria, and the duration of inpatient stay) score. Min 0 p, max > 40 p, higher values worse outcome

SECONDARY OUTCOMES:
Overall Costs of treatment | Costs will be checked at 3 months of follow-up
  Systematic assessment of overall costs

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Acosta, MD PhD, Principal Investigator — Vascular Centre, Malmö, Skåne University Hospital; Julien Hasselmann, MD, Principal Investigator — Vascular Centre, Malmö, Skåne University Hospital
Locations (1):
- Vascular Centre, Malmö, Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Result] Hasselmann J, Bjork J, Svensson-Bjork R, Acosta S. Inguinal Vascular Surgical Wound Protection by Incisional Negative Pressure Wound Therapy: A Randomized Controlled Trial-INVIPS Trial. Ann Surg. 2020 Jan;271(1):48-53. doi: 10.1097/SLA.0000000000003364. PMID 31283565
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Svensson-Bjork R, Hasselmann J, Asciutto G, Zarrouk M, Bjork J, Bilos L, Pirouzram A, Acosta S. Negative Pressure Wound Therapy for the Prevention of Surgical Site Infections Using Fascia Closure After EVAR-A Randomized Trial. World J Surg. 2022 Dec;46(12):3111-3120. doi: 10.1007/s00268-022-06740-5. Epub 2022 Oct 14. PMID 36241857
- [Derived] Rezk F, Astrand H, Acosta S. Incisional negative pressure wound therapy for the prevention of surgical site infection after open lower limb revascularization - Rationale and design of a multi-center randomized controlled trial. Contemp Clin Trials Commun. 2019 Oct 14;16:100469. doi: 10.1016/j.conctc.2019.100469. eCollection 2019 Dec. PMID 31701043
- See also: Study protocol — https://www.scirp.org/journal/paperinformation.aspx?paperid=62452